CLINICAL TRIAL: NCT05206214
Title: Effect of Manual Glide Path Versus Mechanical Glide Path Establishment on Endodontic Postoperative Pain. A Randomized Clinical Trial
Brief Title: Effect of Manual Glide Path Establishment on Endodontic Postoperative Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Elasfouri, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 26-12-2021
Record Dates: First submitted 2021-12-26; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual glide path (Experimental): manual glide path will be established using manual thermal treated stainless-steel files in a watch winding maneuver
  Interventions: Procedure: Manual glide path
- mechanical glide path (Experimental): glide path will be established using rotary Ni-Ti files in a reciprocating maneuver
  Interventions: Procedure: Mechanical glide path

INTERVENTIONS:
Procedure: Manual glide path — manual glide path will be established using manual thermal treated stainless-steel files in a watch winding maneuver. . Coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone.
  Arms: Manual glide path
Procedure: Mechanical glide path — glide path will be established using rotary Ni-Ti files in a reciprocating maneuver. Coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone.
  Arms: mechanical glide path

SUMMARY:
All patients will be treated in a single session approach regardless of the group. All molars will be anesthetized either through infiltration in case of maxillary molars or inferior alveolar nerve block in case of mandibular molars using Octocaine 2% with epinephrine 1: 100,000 (Lidocaine HCl, Novocol Pharmaceutical, Ontario, Canada.). Rubber dam will be applied; and access will be opened using Endo access bur.

In group A manual glide path will be established using manual thermal treated stainless-steel files in a watch winding maneuver. In group B glide path will be established using rotary Ni-Ti files in a reciprocating maneuver. Coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone. Root canals will be copiously irrigated using 10 ml 2.5% sodium hypochlorite NaOCl (Clorox; Egyptian Company for household bleach, Egypt) delivered using 28 Gauge safety Steri Irrigation Tip (DiaDent Group International, Burnaby, BC, Canada) inserted 3 mm below cementoenamel junction. Working length will be determined using electronic apex locator Root ZX II (J. Morita Mfg. Corp, Kyoto, Japan) and confirmed radiographically using parallel technique with receptor holding device. Canals were irrigated again with 10ml 1.5% NaOCl, which was delivered 2mm coronal to apical canal terminus. Irrigation was hydro-dynamically agitated with EndoActivator device (Dentsply Maillefer, Baillagues, Switzerland) using blue tips #30/06 inserted 2mm short of working length for 60 seconds.

DETAILED DESCRIPTION:
All patients will be treated in a single session approach regardless of the group. All molars will be anesthetized either through infiltration in case of maxillary molars or inferior alveolar nerve block in case of mandibular molars using Octocaine 2% with epinephrine 1: 100,000 (Lidocaine HCl, Novocol Pharmaceutical, Ontario, Canada.). Rubber dam will be applied; and access will be opened using Endo access bur.

In group A manual glide path will be established using manual thermal treated stainless-steel files in a watch winding maneuver. In group B glide path will be established using rotary Ni-Ti files in a reciprocating maneuver. Coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone. Root canals will be copiously irrigated using 10 ml 2.5% sodium hypochlorite NaOCl (Clorox; Egyptian Company for household bleach, Egypt) delivered using 28 Gauge safety Steri Irrigation Tip (DiaDent Group International, Burnaby, BC, Canada) inserted 3 mm below cementoenamel junction. Working length will be determined using electronic apex locator Root ZX II (J. Morita Mfg. Corp, Kyoto, Japan) and confirmed radiographically using parallel technique with receptor holding device. Canals were irrigated again with 10ml 1.5% NaOCl, which was delivered 2mm coronal to apical canal terminus. Irrigation was hydro-dynamically agitated with EndoActivator device (Dentsply Maillefer, Baillagues, Switzerland) using blue tips #30/06 inserted 2mm short of working length for 60 seconds. Root canals will be shaped using ProTaper next rotary Ni-Ti files (Dentsply Maillefer, Baillagues, Switzerland). Finally, Root canals will be obturated using cold lateral compaction technique. The molars will be permanently restored using composite resin restoration and will be scheduled for extra coronal restoration.

ELIGIBILITY:
Inclusion Criteria:

* Patient age above 18-70 years old.
* Both males and females will be included.
* All patients are in a good health without systemic condition.
* The offending tooth is a molar.
* The offending molar is indicated for root canal treatment.
* One molar for every patient.
* All patients will sign an informed consent.

Exclusion Criteria:

* 1. The offending tooth has previous attempt of pulp therapy or root canal treatment.
* 2. The patient showing any clinical or radiographic evidence of periapical pathosis.
* 3. Patients received analgesics or systemic antibiotic prior to treatment.

  -.4 Immunocompromised patients.
* 5. Any unknown infectious disease (e.g. HBV, HCV, HIV, or T.B.)
* 6. History of cancer with radio or chemotherapy.
* 7. Offending molar with mobility score ≥2.
* 8. Offending molar with pocket depth ≥6mm.
* 9. Immature molars.
* 10. Nonodontogenic pain.
* 11. Patients with more than one tooth requiring endodontic intervention.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | after 4 hours after root canal treatment
  postoperative pain after root canal treatment using VAS
postoperative pain | after 6hours after root canal treatment
  postoperative pain after root canal treatment using VAS
postoperative pain | after 12hours after root canal treatment
  postoperative pain after root canal treatment using VAS
postoperative pain | after 24hours after root canal treatment
  postoperative pain after root canal treatment using VAS
postoperative pain | after 48 hours after root canal treatment
  postoperative pain after root canal treatment using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Heba A ElAsfouri, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu H, Peng C, Bai Y, Hu X, Wang L, Li C. Shaping ability of ProTaper Universal, WaveOne and ProTaper Next in simulated L-shaped and S-shaped root canals. BMC Oral Health. 2015 Mar 1;15:27. doi: 10.1186/s12903-015-0012-z. PMID 25886847